CLINICAL TRIAL: NCT03093428
Title: A Randomized, Phase II Study Evaluating the Addition of Pembrolizumab (MK-3475) to Radium-223 in Metastatic Castration Resistant Prostate Cancer (mCRPC)
Brief Title: Study Evaluating the Addition of Pembrolizumab to Radium-223 in mCRPC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Atish Choudhury, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-498
Record Dates: First submitted 2017-03-15; First posted 2017-03-28 (Actual); Results first posted 2022-07-20 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radium-223; radium Ra 223 dichloride; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab Plus Radium-223 (Experimental): * Radium-223 will be administered intravenously every 4 weeks at a pre-determined dose
  * Pembrolizumab will be administered intravenously every 3 weeks at a pre-determined dose
  Radium-223 will be halted after 3 doses. Once radiographic progressive disease occurs, the last 3 doses of radium will be given.
  Interventions: Drug: Radium-223; Drug: Pembrolizumab
- Radium-223 (Experimental): - Radium-223 will be administered intravenously every 4 weeks at a pre-determined dose
  Interventions: Drug: Radium-223

INTERVENTIONS:
Drug: Radium-223 — Radium-223 is a calcium mimetic that hones in on bone metastases. It binds to new bone stroma and emits alpha particles, which induce double-stranded DNA breaks that result in tumor cell death.
  Other Names: Xofigo
Drug: Pembrolizumab — Pembrolizumab is a PD-1 inhibitor. Pembrolizumab binds to human PD-1 and blocks the interaction between PD1 and its ligands.
  Other Names: Keytruda
  Arms: Pembrolizumab Plus Radium-223

SUMMARY:
This research study is studying the safety and tolerability of an investigational combination of drugs, radium-223 plus pembrolizumab as a possible treatment for castration-resistant prostate cancer.

The interventions involved in this study are:

* Radium-223
* Pembrolizumab

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has approved radium-223 by itself as a treatment option for the participant's disease.

The FDA has not approved pembrolizumab for the participant's specific disease, but it has been approved for other uses, such as a type of skin cancer called melanoma.

In this research study, the investigators are evaluating the immune response, safety and tolerability of the combination of pembrolizumab (a type of immunotherapy drug) plus radium-223. Pembrolizumab works to block the PD-1 pathway, which plays an important role in lessening the activity of one's immune system to fight cancer. Pembrolizumab is therefore referred to as a PD-1 inhibitor, and acts by stimulating the patient's T cells, which are important immune cells, to attack tumors and treat cancer. Radium-223 targets cancer that exists in the bone directly. Radium-223 binds to minerals in the bone to deliver radiation directly to the cancer that has spread to the bones while limiting damage to the surrounding body tissues. Part of this study is to look at whether the investigators may more effectively control the participant's prostate cancer by combining these drugs. Radium-223 may kill cancer cells and release proteins specific to the tumor. The participant's immune system can then use those proteins to teach the T cells what the cancer looks like, and identify it for attack. Pembrolizumab can increase the number and activity of these immune cells, building a T cell "army" specialized to recognize and attack the cancer. The way these two drugs work on the cancer and the immune system may result in better control of the tumor than just radium-223 alone but needs to be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Castration-resistant prostate cancer requires the following 3 criteria:

  * Progression after surgical castration or on GnRH agonist or antagonist
  * A castrate level of testosterone (<50ng/dL)
  * Prostate cancer progression documented by PSA rise or bone progression according to PCWG2
* There is no limit to number of prior therapies
* Metastatic disease by bone scan
* Age ≥18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Be willing to undergo a core or excisional biopsy of a bone metastasis prior to study drug initiation for tumor tissue. Newly-obtained is defined as a specimen obtained up to 12 weeks (84 days) prior to initiation of treatment on Day 1. Bone biopsy can have been done prior to screening; archival specimens of bone metastasis are permitted if done for other purpose and available.

  --If biopsy is non-diagnostic, patient must undergo repeat biopsy as proof of tumor tissue by pathology review. Proof of tumor specimen is required for eligibility.
* Be willing to undergo a second core or excisional biopsy of a bone metastasis on therapy (approximately after 8 weeks of study therapy or after 2 doses of radium-223 if delays have occurred).
* Demonstrate adequate organ function as defined below, all screening labs for eligibility should be performed within 30 days prior to treatment initiation.
* Hematological

  * Absolute neutrophil count (ANC) ≥ 1,500 /mcL
  * Platelets ≥ 100,000 / mcL
  * Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L; transfusions permitted
* Renal

  --Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤ 1.5 X institutional upper limit of normal (ULN) OR

  ≥30 mL/min for subject with creatinine levels > 1.5 X institutional ULN
* Hepatic

  * Serum total bilirubin ≤ 1.5 X institutional ULN OR Direct bilirubin ≤ institutional ULN for subjects with total bilirubin levels > 1.5 institutional ULN
  * AST (SGOT) and ALT (SGPT) ≤ 2.5 X institutional ULN
  * Albumin > 2.5 mg/dL
* Coagulation

  --International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X institutional ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
  * Activated Partial Thromboplastin Time (aPTT) ≤1.5 X institutional ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
  * Creatinine clearance should be calculated per institutional standard.
* The effects of radium-223 and pembrolizumab on the developing human fetus are unknown. For this reason, men must agree to use adequate contraception. Specifically, they must agree to use a condom (even men with vasectomies) and another effective method of birth control if he is having sex with a woman of childbearing potential or agree to use a condom if he is having sex with a woman who is pregnant while on study drug and for 120 days (4 months) following the last dose of study drug. They must also agree not to donate sperm during the study and for 4 months after receiving the last dose of study drug.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Pathology consistent with majority of specimen having small cell carcinoma of the prostate (prostate cancer with other neuroendocrine features is acceptable).
* Prior treatment with radium-223
* Prior treatment with a PD-1, PD-L1, or PD-L2 blocking therapy
* Evidence of nodal disease greater than or equal to 15 mm in short axis as these findings are concerning for metastases that would not be targeted with radium-223 alone (Arm B). However, lymph nodes with short axis measurements between 1.5-3cm that have not enlarged more than 5mm (to account for reader variability) over the last 6 months and which are not inducing symptoms, causing obstruction, or in the opinion of the investigator pose a risk of impending obstruction of any structures, will be allowed.
* Pulmonary nodules >10 mm

  --Pulmonary nodules >10mm that have been stable for >6 months and are not clearly metastatic disease per the treating investigator are permitted
* Soft tissue components of bone metastases ≥ 1.0 cm in longest axis

  --Soft tissue components of bone metastases < 1.0 cm that have been stable for >6 months (must not have enlarged > 5mm) are permitted
* Soft tissue lesions ≥ 1.0 cm in longest axis

  --Soft tissue lesions < 1.0 cm that have been stable for > 6 months (must not have enlarged > 5mm) are permitted.
* If present, primary disease in the prostate must be stable for > 6 months (defined as no growth > 5mm)
* Evidence of local recurrence in the prostate bed
* Evidence of liver metastases or visceral disease
* Has a diagnosis of immunodeficiency
* Receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., limited low-dose dexamethasone for nausea, multiple doses for contrast allergy) may be enrolled in the study and would not require a 7 day washout.
* Has a known history of active TB (Bacillus Tuberculosis)
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior systemic therapy (exception: GnRH agonist or antagonist) or radiation therapy for prostate cancer within 2 weeks prior to study Day 1. There must be at least a 2 week washout period from last dose of any prior systemic or radiation therapy for prostate cancer prior to Day 1 of study treatment (including nonsteroidal antiandrogens). Screening may commence during this washout window.
* Any patient who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered systemic agent or radiation therapy.

  * Exceptions: Subjects with ≤ Grade 2 neuropathy, hot flashes, or hypertension may qualify for the study if all other eligibility criteria met.
  * Other toxicity or complications that are deemed by the treating investigator as not clinically significant (e.g., urinary incontinence from past prostatectomy)
* Diethylstilbestrol, estrogens, saw palmetto, or other preparations that are known to have possible endocrine effects on prostate cancer that have been started within the past 8 weeks, as they may affect PSA levels or response. These are allowed if the patient has been on a stable dose for at least 8 weeks prior to C1D1.
* Receiving other investigational agents
* History of allergic reactions to compounds with similar biologic or chemical composition to pembrolizumab or Radium-223
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has is planned for curative therapy.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
* Has known history of, or any evidence of active, non-infectious pneumonitis. A history of radiation pneumonitis which is asymptomatic with no signs of active process is allowed.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies). HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with pembrolizumab. In addition, these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA is detected).
* Has received a live vaccine within 30 days of planned start of study therapy.
* Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, severe or unstable angina, myocardial infarction, symptomatic congestive heart failure (defined as New York Heart Association Grade II or greater), arterial or venous thromboembolic events (e.g., pulmonary embolism, cerebrovascular accident including transient ischemic attacks) or clinically significant ventricular arrhythmias within 6 months prior to randomization; or significant vascular disease (e.g., aortic aneurysm, aortic dissection), symptomatic peripheral vascular disease
* Evidence of QTc prolongation as defined as QTcF > 470 ms
* Inability to comply with study and/or follow-up procedures

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2020-04-09 (Actual); Study Completion 2025-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Atish Choudhury, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were enrolled and underwent bone biopsy prior to randomization.
Groups:
- Pembrolizumab Plus Radium-223: * Radium-223 will be administered intravenously every 4 weeks at a pre-determined dose
  * Pembrolizumab will be administered intravenously every 3 weeks at a pre-determined dose
  Radium-223 will be halted after 3 doses. Once radiographic progressive disease occurs, the last 3 doses of radium will be given.
  Radium-223: Radium-223 is a calcium mimetic that hones in on bone metastases. It binds to new bone stroma and emits alpha particles, which induce double-stranded DNA breaks that result in tumor cell death.
  Pembrolizumab: Pembrolizumab is a PD-1 inhibitor. Pembrolizumab binds to human PD-1 and blocks the interaction between PD1 and its ligands.
Period: Overall Study
Arm/Group | Pembrolizumab Plus Radium-223 | Radium-223
Started | 31 | 14
Completed | 12 | 8
Not Completed | 19 | 6
Not completed — Not eligible for treatment | 2 | 1
Not completed — Progression | 14 | 4
Not completed — Death | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Participants who initiated at least one dose of study treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab Plus Radium-223 | Radium-223 | Total
Number analyzed (Participants) | 29 | 13 | 42
Age, Continuous [Median (Full Range); unit: years] | 69 [58 to 79] | 71 [60 to 81] | 70 [58 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 29 | 13 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 27 | 12 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Volume of bone metastases [Count of Participants; unit: Participants]
  < 4 bone metastases | 4 | 1 | 5
  ≥ 4 bone metastases | 25 | 12 | 37
Alkaline phosphatase [Count of Participants; unit: Participants]
  < 220U/L | 21 | 11 | 32
  ≥ 220 U/L | 8 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Increased Immune Cell Infiltration Across Arms
Description: Differences in immune infiltrating cells (CD8+ T-cells and CD4+ T-cells) in bone biopsy specimens were compared from baseline to 8 weeks on study therapy between the treatment arms.
Time Frame: 2 months
Population: Participants who initiated at least one dose of study treatment and available bone biopsy data on baseline and 8-week on treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab Plus Radium-223 | Radium-223
Number analyzed (Participants) | 21 | 5
Participants
  CD4+ T-cell infiltration levels: Increase | 7 | 2
  CD4+ T-cell infiltration levels: No increase | 14 | 3
  CD8+ T-cell infiltration levels: Increase | 3 | 1
  CD8+ T-cell infiltration levels: No increase | 18 | 4

2. Secondary Outcome: Number of Participants With Grade 3 or Higher Treatment Related Adverse Events
Description: Adverse events were assessed using NCI CTCAE (version 4.0). Treatment related adverse events were those that were deemed as "Definitely", "Probably" and "Possibly" related to the study treatment.
Time Frame: Toxicity was assessed every cycle and up to 22.4 months.
Population: Participants who initiated at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab Plus Radium-223 | Radium-223
Number analyzed (Participants) | 29 | 13
Participants | 13 | 5

3. Secondary Outcome: Median Progression-Free Survival
Description: Progression-free survival (PFS) is defined as the time from the first dose of study drug to the earlier of the first documentation of definitive disease progression by RECIST v 1.1 for soft tissue disease and PCWG2 guidelines for bone disease or death due to any cause, or censored at last imaging date.
  Per RECIST, progression is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
  For the bone per PCWG2 criteria, appearance of at least 2 new lesions within 12 weeks and confirmed by a second scan >=6 weeks.
  Median PFS is estimated using Kaplan-Meier method.
Time Frame: Imaging was performed every 12 weeks and up to 25 months.
Population: Participants who initiated at least one dose of study treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab Plus Radium-223 | Radium-223
Number analyzed (Participants) | 29 | 13
Months | 6.1 [2.7 to 10.8] | 5.7 [2.6 to NA] — Not enough subjects had progression or died to estimate the upper confidence limit within follow-up to 25 months.

4. Secondary Outcome: Median Overall Survival
Description: Overall Survival (OS) is defined as the time from randomization (or registration) to death due to any cause, or censored at date last known alive. Median OS is estimated using Kaplan-Meier method.
Time Frame: Participants were followed up for ~36 months.
Population: Participants who initiated at least one dose of study treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab Plus Radium-223 | Radium-223
Number analyzed (Participants) | 29 | 13
Months | 16.9 [12.7 to NA] — Not enough subjects died to estimate the upper confidence limit within follow-up to 30 months. | 16.0 [9.0 to NA] — Not enough subjects died to estimate the upper confidence limit within follow-up to 30 months.

ADVERSE EVENTS:
Time Frame: AE was measured from baseline to end of treatment. Participants were on study up to 35 and 27months for combination and monotherapy arms, respectively.
Description: A serious adverse event is classified using physician's discretion. All adverse events resulting in death, life threatening events, significant disability, prolonged hospitalization, congenital abnormality/birth defect, or new cancer will be considered a serious adverse event.
Arm/Group | Pembrolizumab Plus Radium-223 | Radium-223
All-Cause Mortality (participants affected / at risk) | 15/31 | 7/14
Serious Adverse Events (participants affected / at risk) | 9/31 | 3/14
Other Adverse Events (participants affected / at risk) | 30/31 | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab Plus Radium-223 (N=31) | Radium-223 (N=14)
Abducens nerve disorder (Nervous system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 2 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Oculomotor nerve disorder (Nervous system disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Renal calculi (Renal and urinary disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Stroke (Nervous system disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
White blood cell decreased (Investigations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab Plus Radium-223 (N=31) | Radium-223 (N=14)
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 4 | 0
Alkaline phosphatase increased (Investigations) | 9 | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Anemia (Blood and lymphatic system disorders) | 14 | 4
Anorexia (Metabolism and nutrition disorders) | 8 | 1
Anxiety (Psychiatric disorders) | 7 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 0
Aspartate aminotransferase increased (Investigations) | 11 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 5
Bloating (Gastrointestinal disorders) | 0 | 1
Blood bilirubin increased (Investigations) | 3 | 0
Blurred vision (Eye disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Breast pain (Reproductive system and breast disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 0
CD4 lymphocytes decreased (Investigations) | 1 | 2
Chills (General disorders) | 0 | 1
Cholesterol high (Investigations) | 1 | 0
Concentration impairment (Nervous system disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 12 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Creatinine increased (Investigations) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Depression (Psychiatric disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 11 | 5
Dizziness (Nervous system disorders) | 3 | 0
Dry eye (Eye disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0
Dysgeusia (Nervous system disorders) | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 | 1
Edema limbs (General disorders) | 4 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 2 | 0
Eye disorders - Other, specify (Eye disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Fatigue (General disorders) | 26 | 10
Fever (General disorders) | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Flu like symptoms (General disorders) | 2 | 0
Fracture (Injury, poisoning and procedural complications) | 3 | 0
Gait disturbance (General disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 1
Gynecomastia (Reproductive system and breast disorders) | 1 | 2
Headache (Nervous system disorders) | 4 | 1
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Hematoma (Vascular disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Hot flashes (Vascular disorders) | 13 | 5
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 3
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 7 | 6
Hyperthyroidism (Endocrine disorders) | 4 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 4 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 0
Hypothyroidism (Endocrine disorders) | 10 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Injection site reaction (General disorders) | 1 | 0
INR increased (Investigations) | 1 | 0
Insomnia (Psychiatric disorders) | 4 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Libido decreased (Psychiatric disorders) | 2 | 0
Localized edema (General disorders) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 | 0
Middle ear inflammation (Ear and labyrinth disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 14 | 3
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 5 | 1
Non-cardiac chest pain (General disorders) | 2 | 0
Pain (General disorders) | 13 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 1
Paresthesia (Nervous system disorders) | 3 | 0
Periodontal disease (Gastrointestinal disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 2
Personality change (Psychiatric disorders) | 1 | 0
Platelet count decreased (Investigations) | 7 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 1
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 1
Seizure (Nervous system disorders) | 1 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 | 0
Skin infection (Infections and infestations) | 4 | 0
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 2
Thromboembolic event (Vascular disorders) | 4 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0
Urinary frequency (Renal and urinary disorders) | 7 | 4
Urinary incontinence (Renal and urinary disorders) | 5 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Weight loss (Investigations) | 2 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
White blood cell decreased (Investigations) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT03093428/Prot_SAP_000.pdf